CLINICAL TRIAL: NCT02909478
Title: Steroid-free Regimen With Aprepitant in Preventing Chemotherapy-induced Nausea and Vomiting in Patients With Colorectal Cancer Receiving FOLFOX Chemotherapy: a Randomized Phase 3 Trial
Brief Title: Aprepitant Without Steroid in Preventing Chemotherapy-induced Nausea and Vomiting in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GIHSYSU12
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Colorectal Cancer
MeSH Terms: conditions — Vomiting; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprepitant arm (Experimental): Aprepitant + Tropisetron
  Interventions: Drug: Aprepitant+Tropisetron
- Control arm (Active Comparator): Dexamethasone+ Tropisetron
  Interventions: Drug: Dexamethasone+Tropisetron

INTERVENTIONS:
Drug: Aprepitant+Tropisetron — Patients will receive the chemotherapy drugs oxaliplatin,leucovorin and 5-fluorouracil as well as the following antiemetic drugs:
  aprepitant (125 mg orally on day 1 and 80 mg orally on days 2 and 3) plus Tropisetron (5mg IV of day1)
  Arms: Aprepitant arm
Drug: Dexamethasone+Tropisetron — Patients will receive the chemotherapy drugs oxaliplatin, leucovorin and 5-fluorouracil as well as the following antiemetic drugs:
  Dexamethasone (10 mg IV on day 1 and 5 mg IV days 2, 3) plus Tropisetron (5mg IV of day1)
  Arms: Control arm

SUMMARY:
Addition of aprepitant, an NK1 receptor antagonist to a 5-HT3 receptor antagonist and dexamethasone regimen was shown to be effective for prevention of chemotherapy-induced nausea and vomiting (CINV) with moderately emetogenic chemotherapy (MEC). Little is known about the efficacy of aprepitant when used without dexamethasone. Dexamethasone is widely used to prevent both acute and delayed nausea and vomiting induced by chemotherapy. However, multi-period use of dexamethasone could be associated with side effect, such as hyperglycemia, dyspepsia and insomnia. This randomized phase III trial studies antiemetic therapy with aprepitant and tropisetron to see how well they work compared to dexamethasone plus tropisetron in preventing chemotherapy-induced nausea and vomiting in patients with colorectal cancer receiving FOLFOX(oxaliplatin, leuvovorin and 5-fluorouracil) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer
* No prior chemotherapy and scheduled to receive FOLFOX chemotherapy (oxaliplatin,leucovorin and 5-fluorouracil)
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Laboratory index: Hemoglobin ≥ 90 g/L (No blood transfusion within 14 days), Absolute Neutrophil Count ≥ 1.5×10^9/L, Platelet Count ≥ 75×10^9/L, Serum Bilirubin ≤ 1.5×ULN, ALT and AST ≤ 3.0×ULN (without liver metastases), ALT and AST ≤ 5.0×ULN (with liver metastases), Serum Creatinine ≤ 1×ULN, Endogenous Creatinine Clearance>60ml/min
* Be able to read, understand and complete the questionnaire and diary
* Be able to understand the study procedures and sign informed consent.

Exclusion Criteria:

* Treatment with any other study medicine within 4 weeks before enrollment.
* Nausea or vomiting ≤ 24 hours prior to registration
* Ongoing emesis due to obstruction of digestive tract
* Concurrent use of olanzapine, phenothiazine or amifostine
* Female with pregnancy or lactation
* Severe cognitive compromise
* Known history of CNS disease (e.g. brain metastases, seizure disorder)
* Concurrent abdominal radiotherapy
* Chronic alcoholism
* Known hypersensitivity to aprepitant, tropisetron, or dexamethasone.
* Known cardiac arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within the previous six months.
* History of uncontrolled diabetes mellitus
* Serious or uncontroled infection
* Known active HIV, viral hepatitis or tuberculosis infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Complete response | Day 1 to Day 5 after chemotherapy
  No emetic episodes and no use of rescue medication

SECONDARY OUTCOMES:
Nausea score | Day 1 to Day 5 after chemotherapy
  Nausea scores measured by the Nausea and Vomiting Daily Diary/Questionnaire
Time to First Vomiting Episode or Use of Rescue Medication | Day 1 to Day 5 after chemotherapy
Frequency of rescue medication | Day 1 to Day 5 after chemotherapy
  Patients were asked to record daily number of extra nausea/vomiting pills taken because they developed nausea/vomiting in the following categories: None, One, Two, More than two in Nausea and Vomiting Daily Diary Questionnaire
Complete response in the acute phase (0-24 hours) | 0 to 24 hours after chemotherapy
  No emetic episodes and no use of rescue medication in the acute phase (0-24 h)
Complete response in the delay phase (25 hours-120 hours) | Day 2 to Day 5 (25 hours-120 hours) after chemotherapy
  No emetic episodes and no use of rescue medication in the delay phase

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Cheng Y, Wu Z, Shi L, Shen C, Zhang J, Hu H, Li W, Cai Y, Xie X, Ling J, Zheng Q, Deng Y. Aprepitant plus palonosetron versus dexamethasone plus palonosetron in preventing chemotherapy-induced nausea and vomiting in patients with moderate-emetogenic chemotherapy: A randomized, open-label, phase 3 trial. EClinicalMedicine. 2022 Jun 3;49:101480. doi: 10.1016/j.eclinm.2022.101480. eCollection 2022 Jul. PMID 35747189